CLINICAL TRIAL: NCT06464276
Title: Effectiveness and Tolerability of Trimetazidine 80mg Once Daily in Patients With Chronic Coronary Syndrome: The V-GOOD Observational Study
Brief Title: Effectiveness and Tolerability of Trimetazidine 80mg Once Daily in Patients With Chronic Coronary Syndrome: The V-GOOD Study
Acronym: V-GOOD
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Brazil (Other Government)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Luis Henrique W Gowdak, MD, PhD, Principal Investigator, Ministry of Health, Brazil
Other Study IDs: 49351321.8.0000.0068
Record Dates: First submitted 2024-06-07; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Chronic Coronary Syndrome; Stable Angina
Keywords: Trimetazidine; Angina Pectoris; Stable Angina; Medication Adherence
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed Chronic Coronary Syndrome and persistent stable angina.: Patients with confirmed Chronic Coronary Syndrome and persistent stable angina will be observed without any intervention, and the study will follow them for 3 months while they are treated with Trimetazidine 80 mg OD.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The objective of this non-interventional multicentric study (NIS) is to investigate the efficacy and tolerability of treatment with Vastarel Caps LP® in symptomatic patients with angina over 3 months under conditions of daily practice. The main questions it aims to answer are data collection on antianginal efficacy, symptom class, adherence, and overall tolerability in patients treated with Vastarel Caps LP®.

Patients diagnosed with chronic coronary syndrome and persistent stable angina, for whom the cardiologist chose to prescribe Trimetazidine 80mg once daily, were included in the study. Clinical information was collected in three distinct visits at baseline (V1), 1 month (V2), and 3 months (V3). During these visits, cardiologists collected the following variables based on a weekly occurrence: number of angina crises, short-acting nitrates (SAN) consumption, Canadian Cardiovascular Society (CCS) classification, level of self-reported daily physical activity, adherence, and tolerability to the treatment. Physical activity was measured using a scale from 1 to 10 (1 = no limitations, 5 = moderate limitations, and 10 = very marked limitations). Adherence was assessed by a previously validated six-item questionnaire. Assessment of therapy efficacy and tolerability were rated by the physician as "very satisfactory", "satisfactory", "not sufficiently satisfactory", and "unsatisfactory".

DETAILED DESCRIPTION:
Patients must be informed about their participation in this study and the transfer of their clinical data outside the research center to statistical data analysts. The patient consent form must be obtained in writing. Patients diagnosed with chronic coronary syndrome and persistent stable angina, for whom the cardiologist chose to prescribe Trimetazidine 80mg once daily, were included in the study. Clinical information was collected in three distinct visits at baseline (V1), 1 month (V2), and 3 months (V3). During these visits, cardiologists collected the following variables based on a weekly occurrence: number of angina crises, short-acting nitrates (SAN) consumption, Canadian Cardiovascular Society (CCS) classification, level of self-reported daily physical activity, adherence, and tolerability to the treatment. Physical activity was measured using a scale from 1 to 10 (1 = no limitations, 5 = moderate limitations, and 10 = very marked limitations). Adherence was assessed by a previously validated six-item questionnaire. Assessment of therapy efficacy and tolerability were rated by the physician as "very satisfactory", "satisfactory", "not sufficiently satisfactory", and "unsatisfactory".

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Chronic Coronary Syndrome and persistent stable angina;
* Patients who are going to start using Vastarel Caps LP® as per their doctor's recommendation.

Exclusion Criteria:

* Hypersensitivity to the active ingredient or any of the excipients listed in Vastarel Caps LP®;
* Parkinson's disease, Parkinson's symptoms, tremors, restless leg syndrome, and other related movement disorders;
* Severe renal impairment (creatinine clearance <30 mL/min);
* Moderate renal impairment (creatinine clearance [30-60] mL/min).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stable chronic angina who are considered eligible for treatment with Vastarel Caps LP® by their physicians are suitable for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of Vastarel Caps LP® therapy on frequency of angina episodes. | 30 days (V2), 90 days (V3)
  Assessment of the effect of Vastarel Caps LP® therapy on changing the number of angina attacks at 30 and 90 days, as reported by the patient.
Effect of Vastarel Caps LP® therapy on the use of sublingual nitrates. | 30 days (V2), 90 days (V3)
  Assessment of the effect of Vastarel Caps LP® therapy on the alteration of sublingual nitrates consumption at 30 days and 90 days.
Effect of Vastarel Caps LP® therapy on symptom class (CCS class). | 30 days (V2), 90 days (V3)
  Assessing the impact of Vastarel Caps LP® therapy on modifying symptom classification using the CCS class at 30 and 90 days.
Effect of Vastarel Caps LP® therapy on daily activity. | 30 days (V2), 90 days (V3)
  Assessment of the impact of Vastarel Caps LP® therapy on adjusting the daily activity threshold at 30 and 90 days, utilizing the Functional Assessment Scale to be answered by the patient.
Influence of Vastarel Caps LP® therapy on patient adherence. | 30 days (V2), 90 days (V3)
  Assessment of the impact of Vastarel Caps LP® therapy on enhancing patient adherence at 30 and 90 days, through the following questions: This morning, did you forget to take Vastarel Caps LP? Yes or No, Since our last appointment, have you taken Vastarel Caps LP after the usual time? Yes or No and Since our last appointment, have you ever forgotten to take Vastarel Caps LP? Yes or No.

SECONDARY OUTCOMES:
Overall tolerability and adverse events (AE)/adverse drug reactions (ADR) in Vastarel Caps LP® therapy | 30 days (V2), 90 days (V3)
  Assessment of the effect of Vastarel Caps LP® therapy on overall patient tolerability and the occurrence of adverse events (AE)/adverse drug reactions (ADR), as reported by the patient through the following question: "How do you assess the overall tolerability of Vastarel Caps LP therapy in this patient? Very satisfactory, Satisfactory, Not satisfactory enough, or Unsatisfactory."
Overall assessment by the physician of the efficacy of Vastarel Caps LP® therapy in symptomatic patients with angina. | 30 days (V2), 90 days (V3)
  Assessment of the efficacy of Vastarel Caps LP® therapy based on the physician's overall evaluation through the following question: "How do you assess the overall effectiveness of Vastarel Caps LP therapy in this patient? Very satisfactory, Satisfactory, Not satisfactory enough, or Unsatisfactory."
Association of Vastarel Caps LP® efficacy according to the time since the patient's last revascularization. | 30 days (V2), 90 days (V3)
  Assessment of the relationship between the time elapsed since the last surgical intervention to enhance blood flow in the coronary arteries and the effectiveness of Vastarel treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luis H Gowdak, PhD, Principal Investigator — InCor Heart Institute
Locations (1):
- InCor Heart Institute, São Paulo, Brazil

REFERENCES:
- [Derived] Gowdak LHW, Dourado PMM, Precoma DB, de Oliviera Lopes Dusilek C, da Silva FM, Yugar-Toledo JC, Pena FM, de Almeida Gomes DA, do Espirito Santo Cestario E, Guimaraes OR Jr, Filho CRH, de Almeida CF, de Souza Brito F, Martins GF, Ferreira VRR, Flores MC, da Silva ML; V-GOOD Investigators. Effectiveness and Tolerability of Trimetazidine 80 mg Once Daily in Patients with Chronic Coronary Syndrome in Brazil: The V-GOOD Observational Study. Cardiol Ther. 2025 Jun;14(2):249-265. doi: 10.1007/s40119-025-00405-9. Epub 2025 Apr 29. PMID 40299195